CLINICAL TRIAL: NCT05645718
Title: Phase II Study of Pedi-cRIB: Mini-Hyper-CVD With Condensed Rituximab, Inotuzumab Ozogamicin and Blinatumomab (cRIB) for Relapsed Therapy for Pediatric With B-Cell Lineage Acute Lymphocytic Leukemia
Brief Title: Study of Pedi-cRIB: Mini-Hyper-CVD With Condensed Rituximab, Inotuzumab Ozogamicin and Blinatumomab (cRIB) for Relapsed Therapy for Pediatric With B-Cell Lineage Acute Lymphocytic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0312; NCI-2022-10168 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-11-29; First posted 2022-12-09 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia | interventions — Cyclophosphamide; Vincristine; blinatumomab; Methotrexate; Cytarabine; Mercaptopurine; Prednisone; pegfilgrastim; pegylated granulocyte colony-stimulating factor, human; Inotuzumab Ozogamicin; Rituximab; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Leukemia CNS1 or 2 (Experimental): Each study block, or cycle, is 28 days. Between every cycle below, Participants will have a 7-day rest period in which no study drug is given.
  Interventions: Drug: Cyclophosphamide; Drug: Vincristine; Drug: Blinatumomab; Drug: Methotrexate; Drug: Cytarabine; Drug: Mercaptopurine; Drug: Prednisone; Drug: Pegfilgrastim; Drug: Inotuzumab ozogamicin; Drug: Rituximab; Drug: Dexamethasone
- Leukemia CNS 3 (Experimental): Each study block, or cycle, is 28 days. Between every cycle below, Participants will have a 7-day rest period in which no study drug is given.
  Interventions: Drug: Cyclophosphamide; Drug: Vincristine; Drug: Blinatumomab; Drug: Methotrexate; Drug: Cytarabine; Drug: Mercaptopurine; Drug: Prednisone; Drug: Pegfilgrastim; Drug: Inotuzumab ozogamicin; Drug: Rituximab; Drug: Dexamethasone

INTERVENTIONS:
Drug: Cyclophosphamide — Given by (IV) vein
  Other Names: Cytoxan®; Neosar®
Drug: Vincristine — Given by (IV) vein
Drug: Blinatumomab — Given by (IV) vein
Drug: Methotrexate — Given by (IV) vein
Drug: Cytarabine — Given by (IV) vein
  Other Names: Ara-C; Cytosar®; DepoCyt™; Cytosine arabinosine hydrochloride
Drug: Mercaptopurine — Given by (IV) vein
  Other Names: 6-mercaptopurine; Purinethol®; 6-MP
Drug: Prednisone — Given by PO
Drug: Pegfilgrastim — Given by (IV) vein
  Other Names: NeulastaTM; PEG-G-CSF
Drug: Inotuzumab ozogamicin — Given by (IV) vein
  Other Names: CMC-544
Drug: Rituximab — Given by (IV) vein
  Other Names: Rituxan
Drug: Dexamethasone — Given by (IV) vein
  Other Names: Decadron

SUMMARY:
To learn if cyclophosphamide, vincristine, and dexamethasone (called mini hyper-CVD) in combination with intrathecal (delivered into the spine) chemotherapy (methotrexate, hydrocortisone, cytarabine) and compressed rituximab, blinatumomab, and inotuzumab ozogamicin (called cRIB) can help to control the disease.

DETAILED DESCRIPTION:
Primary Objective:

--To evaluate the clinical efficacy of the sequential combination of mini-hyper-CVD with inotuzumab ozogamicin and blinatumomab and rituximab in relapsed B-cell acute lymphoblastic leukemia (ALL) patients, based upon the complete response rate (CR).

Secondary Objectives:

* To summarize efficacy per response rate, overall survival (OS), event free survival (EFS), and minimal residual disease (MRD) negativity rate.
* To evaluate the safety of this combination.

Exploratory Objectives:

--To summarize associations between genomic alterations in ALL (current biomarker expression of the disease) with relation to the incidence of transition to HSCT in patients with PR or stable disease (SD) after the induction cycle(s).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric, adolescent, or young adult patients with B-ALL as per NCCN v2.2021 and WHO classification in relapse or primary refractory and, either/both of the following: • Unable to receive anthracyclines (see section 3.1.8) or is PEG-asparaginase intolerant.

  * For leukemia: Patients must have ≥ 5% blasts expressing CD19 and CD22 in the bone marrow as assessed by morphology or flow cytometry. However, if an adequate bone marrow sample cannot be obtained, patients may be enrolled if there is unequivocal evidence of leukemia with ≥ 5% blasts in the peripheral blood.
  * If patient does not have CD20, they can still be enrolled but will not receive rituximab.
* Performance status: Lansky ≥ 50 for patients who are ≤ 16 years old and Karnofsky ≥ 50% for patients who are > 16 years old.
* Patients with asymptomatic CNS leukemia are eligible (see also Exclusion Criterion 3.2.2.)
* Age > = 1 years of age and less than 25 years of age.
* The following baseline laboratory data:

  * Total serum bilirubin ≤1.5x upper limit of normal (ULN). Patients with known Gilbert's syndrome may have a total bilirubin up to ≤3 x ULN.
  * Adequate renal function per age51 unless related to the disease. Estimated glomerular filtration rate ≥ 60 mL/min/1.73 m2 based on local institutional practice for age-appropriate determination (eg, Schwartz formula for pediatric patients or Cockcroft Gault formula for adults).
  * Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤3 x ULN; ≤5 x ULN in case of suspected leukemic liver involvement
* Females of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test result within 14 days prior to the first dose of study drugs and must agree to use one of the following effective contraception methods during the study and 30 days after the last treatment and 8 months after the last dose of inotuzumab and 12 months after the last dose of rituximab. Effective methods of birth control include:

  * Birth control pills, shots, implants (placed under the skin by a health care provider) or patches (placed on the skin)
  * Intrauterine devices (IUDs)
  * Condom or occlusive cap (diaphragm or cervical/vault caps) used with Spermicide
  * Abstinence
* Males need to inform the doctor right away if the partner becomes pregnant or suspects pregnancy. While in this study and for 30 days after the last treatment the patient should not donate sperm for the purposes of reproduction. He will need to use a condom while in this study and for 30 days after the last treatment and 5 months after the last dose of inotuzumab.
* Patients with cardiac disease, include but not limited to: (Left ventricular ejection fraction (EF) < 50% (as determined by the Biplane Simpson method) (but not per exclusion criteria 3.2.3.1), or who have received >450mg/m2 of doxorubicin and cannot receive anthracyclines.

Exclusion Criteria:

* Past or current history of a secondary or other primary tumor or a chronic myeloid leukemia (CML) blast crisis with exception of:

  * Curatively treated non-melanomatous skin cancer
  * Other primary solid tumor treated with curative intent and no known active disease present and no treatment administered during the last 2 years
* Presence of clinically significant uncontrolled CNS pathology such as epilepsy, childhood seizure, paresis, aphasia, stroke, severe brain injuries, organic brain syndrome, or psychosis. Presence of the following are allowed: headaches, vomiting, nerve palsy
* Medical history of cardiovascular disease such as:

  ° Clinically significant cardiac disease including congestive heart failure (NYHA class III or IV) or arrhythmia or conduction abnormality requiring medication
* Patients with uncontrolled, active infections (viral, bacterial, or fungal). Infections controlled on concurrent anti-microbial agents are acceptable, and anti-microbial prophylaxis per institutional guidelines are acceptable.
* Known active hepatitis B or C infection or known seropositivity for HIV.
* Patients with liver cirrhosis or other serious active liver disease or with suspected active alcohol abuse.
* Active acute/chronic Graft-versus-Host Disease (GvHD) requiring systemic treatment; or receiving immunosuppression for GvHD prophylaxis within 2 weeks from the start of study therapy.
* If patient has not recovered (as deemed by the investigator) from previous chemotherapy, surgery, radiation before the start of study drugs.

  ° To reduce the circulating blast count or palliation, the following are allowed prior to starting: Single dose intravenous cytarabine, steroids or hydroxyurea. No washout necessary for these agents.
* Females who are pregnant or lactating.
* Male or female subjects of childbearing potential, unwilling to use an approved, effective means of contraception in accordance with institution's standards.
* Other severe, uncontrolled acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated Protocol 2022-0312 V3 Dated 11/9/2023 Property of Leukemia at MD Anderson 17 with study participation or investigational product administration or may interfere with the interpretation of study results and/or would make the patient inappropriate for enrollment into this study.
* Patients with Trisomy 21, or bone marrow failure syndromes are not eligible.
* Prior history of allergic reaction to any of the agents.
* Patients who are unable or unwilling to comply with all study requirements for clinical visits, examinations, tests, and procedures.
* Patients may be excluded if they are currently enrolled in another ongoing clinical trial with investigational products

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: David McCall, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org